CLINICAL TRIAL: NCT00973544
Title: Complications of Breast Reconstruction With Silicone Prosthesis in Relation to Closed Suction Drains
Brief Title: Do Closed Suction Drains Affect the Complications Rate of Breast Reconstruction With Silicone Prosthesis?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Eyal Winkler, MD, Plastic & Reconstructive Department, Sheba Medical Center, Israel
Other Study IDs: SHEBA -08-5530 -EW- CTIL
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Breast Reconstruction
Keywords: breast reconstruction complications; drains; silicone implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cultures of fluids from drain
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: drains would be removed when daily discharge will be below 20 cc for 2 consecutive days
  Interventions: Other: Cultures taken from the drain discharge
- study: drains will be removed on post operative day (POD) 10
  Interventions: Other: Cultures taken from the drain discharge

INTERVENTIONS:
Other: Cultures taken from the drain discharge — Cultures will be taken from drain's fluids discharge in Post Operative Day 4,8,10,12. When drain is removed cultures of the drain tip are taken. Clinical signs of surgical signs infections will be observed.

SUMMARY:
The purpose of this study is to describe the relations between closed suction drains placement in breast reconstructions procedures with silicone prothesis to the development of local wound complications (seroma, hematoma, infections).

DETAILED DESCRIPTION:
Breast reconstruction with silicone prosthesis can be divided into two groups: immediate and late reconstructions. The complications rates reported in the literature are around 30% for delayed reconstructions and 50% for immediate reconstructions. The estimated surgical site infection rate is approximately 7% and seroma formation rate is approximately 1.2%.

In many of the procedures closed suction drains are left for fluid drainage, in order to reduce seroma formation. Still, the timing of drains' removal is controversial. Our aim in this study is to describe the relation between the placement of closed suction drains, the timing for their removal, and immediate post operative complications.

Patients that underwent breast reconstruction with silicone prosthesis and in which drains will be left in the surgical field would be randomly assigned into two groups: a control group, in which drains will be removed when the daily discharge will be below 20 cc for two consecutive days and the study group, in which drains will be removed on post operative day (POD) 10. All patients will receive the same antibiotic prophylaxis regimen. Cultures will be taken from fluid discharge POD 4,8,10 and 12. The incidence of local wound complications such as infection, seroma, hematoma and skin necrosis was record and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent immediate or late breast reconstruction with silicone prosthesis (expanders/implants)and in which closed suction drains were left in the operating field according to the decision of the operating surgeon.
* signature of informed consent form

Exclusion Criteria:

* age under 18
* breast reconstruction without prosthesis
* Breast reconstruction without the use of drains
* Active infection during time of surgery in surgical site
* Coagulation disease
* Psychiatric illness
* Immune disease
* Lack of communication or language problems
* Foreign residents, not Israeli citizens
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent breast reconstruction with silicone prosthesis and in which drains were left in the surgical field. patients will signed an informed consent form
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09